CLINICAL TRIAL: NCT06554665
Title: Powering Up Stroke Rehabilitation Through High-Intensity Interval Training
Brief Title: Powering Up Stroke Rehabilitation Through HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20230720002
Record Dates: First submitted 2024-07-30; First posted 2024-08-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-intensity interval training (Experimental): The HIIT session will consist of a 3-minute warm-up, a 20-minute main exercise, and a 2-minute cool-down. The main exercise for HIIT will include ten high-intensity intervals, interspersed with ten low-intensity intervals.
  Interventions: Behavioral: High-intensity Interval Training
- Moderate-intensity continuous training (Active Comparator): The MICT session will consist of a 3-minute warm-up, a main exercise that is isoenergetic with the HIIT session (lasting approximately 30 minutes), and a 2-minute cool-down. The intensity during the main exercise for MICT will remain constant throughout the session.
  Interventions: Behavioral: Moderate-Intensity Continuous Training
- Stretching (Active Comparator): The stretching group will receive 25 minutes of whole-body stretching.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: High-intensity Interval Training — There will be three sessions per week for 12 consecutive weeks, totaling 36 training sessions.
  Arms: High-intensity interval training
Behavioral: Moderate-Intensity Continuous Training — There will be three sessions per week for 12 consecutive weeks, totaling 36 training sessions.
  Arms: Moderate-intensity continuous training
Behavioral: Stretching — There will be three sessions per week for 12 consecutive weeks, totaling 36 training sessions.
  Arms: Stretching

SUMMARY:
Objectives: To investigate the effects of high-intensity interval training (HIIT) on musculoskeletal fitness in chronic stroke survivors.

Hypothesis to be tested: HIIT, performed on a recumbent stepper, will significantly enhance muscle power in chronic stroke survivors when compared with moderate-intensity continuous training (MICT) Design and subjects: Assessor-blinded, stratified, randomised, placebo-controlled clinical trial involving eligible 66 chronic stroke survivors.

Interventions: Participants will be randomly allocated to one of three groups: the HIIT group, the MICT group, or a stretching group (active control). Each group will attend sessions three times per week for 12 consecutive weeks, totaling 36 training sessions.

Main outcome measures: Assessments will be conducted at baseline, at mid-term of the intervention (week 6), at the end of the intervention (week 12), and at a 12-week follow-up (week 24). The primary outcome measure will be muscle power. Secondary outcome measures will include muscle strength, body composition, biomarkers, motor function, balance function, cardiorespiratory response, and psychosocial response.

ELIGIBILITY:
Inclusion criteria:

* Men and postmenopausal women aged 50-80 years
* 1-5 years following the first-ever stroke confirmed by magnetic resonance imaging or computed tomography
* Able to walk 10 meters independently with or without a walking aid
* Class I or II according to the New York Heart Association Functional Classification (no limitation or slight limitation of physical activity due to symptoms during ordinary physical activity)

Exclusion criteria:

* Presence of other neurological comorbidities, significant liver or renal diseases, thyroid or parathyroid diseases, rheumatoid arthritis, or a fracture within the past 6 months
* Undergoing osteoporosis treatments within the past 3 years, use of oral corticosteroids for more than 3 months within the past year, or botulinum toxin injections in the paretic lower limb within the past 6 months
* Participation in ongoing stroke rehabilitation services or structured exercise programme
* Cognitive or communication issues that could limit the ability to follow instructions
* Contraindications to HIIT, graded exercise testing, or failure to pass medical clearance from a specialist

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Muscle Power at Week 12 | Baseline and Week 12
  Muscle power (watt) of knee extensors on both the paretic and nonparetic sides will be measured using the isokinetic dynamometer.
  Change=(Week 12 Level - Baseline Level)

SECONDARY OUTCOMES:
Change from Baseline in Muscle Power at Week 24 | Baseline and Week 24
  Muscle power (watt) of knee extensors on both the paretic and nonparetic sides will be measured using the isokinetic dynamometer. Change=(Week 24 Level - Baseline Level)
Change from Baseline in Muscle Strength (Nm) at Week 12 | Baseline and Week 12
  Muscle strength (Nm) of knee extensors on both the paretic and nonparetic sides will be measured using the isokinetic dynamometer.
  Change=(Week 12 Level - Baseline Level)
Change from Baseline in Muscle Strength (Nm) at Week 24 | Baseline and Week 24
  Muscle strength (Nm) of knee extensors on both the paretic and nonparetic sides will be measured using the isokinetic dynamometer.
  Change=(Week 24 Level - Baseline Level)
Change from Baseline in Muscle Strength (kg) at Week 12 | Baseline and Week 12
  Handgrip strength (kg) on both sides will be measured using a handheld dynamometer.
  Change=(Week 12 Level - Baseline Level)
Change from Baseline in Muscle Strength (kg) at Week 24 | Baseline and Week 24
  Handgrip strength (kg) on both sides will be measured using a handheld dynamometer.
  Change=(Week 24 Level - Baseline Level)
Change from Baseline in Body Composition (kg) at Week 12 | Baseline and Week 12
  Whole-body skeletal muscle mass (kg), bone mineral content (kg), fat mass (kg), and segmental lean mass (kg) will be measured using bioelectrical impedance analysis (BIA).
  Change=(Week 12 Level - Baseline Level)
Change from Baseline in Body Composition (kg) at Week 24 | Baseline and Week 24
  Whole-body skeletal muscle mass (kg), bone mineral content (kg), fat mass (kg), and segmental lean mass (kg) will be measured using bioelectrical impedance analysis (BIA).
  Change=(Week 24 Level - Baseline Level)
Change from Baseline in Body Composition (%) at Week 12 | Baseline and Week 12
  Body fat percentage (%) will be measured using bioelectrical impedance analysis (BIA).
  Change=(Week 12 Level - Baseline Level)
Change from Baseline in Body Composition (%) at Week 24 | Baseline and Week 24
  Body fat percentage (%) will be measured using bioelectrical impedance analysis (BIA).
  Change=(Week 24 Level - Baseline Level)
Change from Baseline in Biomarkers at Week 12 | Baseline and Week 12
  Volume-corrected serum concentration (mg/dL) of myokines, bone markers, pro-inflammatory markers, biomarkers of oxidative stress will be measured using enzyme-linked immunosorbent assay (ELISA) kits.
  Change=(Week 12 Level - Baseline Level)
Change from Baseline in Biomarkers at Week 6 | Baseline and Week 6
  Volume-corrected serum concentration (mg/dL) of myokines, bone markers, pro-inflammatory markers, biomarkers of oxidative stress will be measured using enzyme-linked immunosorbent assay (ELISA) kits.
  Change=(Week 6 Level - Baseline Level)
Change from Baseline in Motor Function at Week 12 | Baseline and Week 12
  Fugl-Meyer Motor Assessment (FMA) will be used to assess the degree of motor recovery of the hemiparetic upper (range: 0-66) and lower limbs (range: 0-34). Higher scores are indicative of better motor recovery. Short Physical Performance Battery (SPPB) will be used to assess the physical performance, including 5-times sit-to-stand, balance tests (side-by-side-stand, semi-tandem stand, and tandem stand), and gait speed.
  Change=(Week 12 Score- Baseline Score)
Change from Baseline in Motor Function at Week 24 | Baseline and Week 24
  Fugl-Meyer Motor Assessment (FMA) will be used to assess the degree of motor recovery of the hemiparetic upper (range: 0-66) and lower limbs (range: 0-34). Higher scores are indicative of better motor recovery. Short Physical Performance Battery (SPPB) will be used to assess the physical performance, including 5-times sit-to-stand, balance tests (side-by-side-stand, semi-tandem stand, and tandem stand), and gait speed.
  Change=(Week 24 Score- Baseline Score)
Change from Baseline in Motor Function (meters) at Week 12 | Baseline and Week 12
  The 6-minute walk test (6MWT) will be used to measure walking endurance and capacity. The total distance walked in meters during the test will be recorded.
  Change=(Week 12 distance - Baseline distance)
Change from Baseline in Motor Function (meters) at Week 24 | Baseline and Week 24
  The 6-minute walk test (6MWT) will be used to measure walking endurance and capacity. The total distance walked in meters during the test will be recorded.
  Change=(Week 24 distance - Baseline distance)
Change from Baseline in Balance Function at Week 12 | Baseline and Week 12
  Balance performance will be assessed using the Mini Balance Evaluation Systems Test (range: 0-28). Higher scores are indicative of better balance performance. Fear of falling will be assessed using the Chinese version of the Activities-Specific Balance Confidence Scale (range: 0-100). Higher scores are indicative of higher balance confidence.
  Change=(Week 12 Score- Baseline Score)
Change from Baseline in Balance Function at Week 24 | Baseline and Week 24
  Balance performance will be assessed using the Mini Balance Evaluation Systems Test (range: 0-28). Higher scores are indicative of better balance performance. Fear of falling will be assessed using the Chinese version of the Activities-Specific Balance Confidence Scale (range: 0-100). Higher scores are indicative of higher balance confidence.
  Change=(Week 24 Score- Baseline Score)
Change from Baseline in Cardiopulmonary Response at Week 12 | Baseline and Week 12
  Peak oxygen uptake (VO2peak) will be measured using a graded exercise test (GXT). The GXT will be conducted following a well-validated protocol that on a whole-body recumbent stepper to assess cardiopulmonary function in stroke patients.
  Change=(Week 12 VO2peak - Baseline VO2peak)
Change from Baseline in Cardiopulmonary Response at Week 24 | Baseline and Week 24
  Peak oxygen uptake (VO2peak) will be measured using a graded exercise test (GXT). The GXT will be conducted following a well-validated protocol that on a whole-body recumbent stepper to assess cardiopulmonary function in stroke patients.
  Change=(Week 24 VO2peak - Baseline VO2peak)
Change from Baseline in Psychosocial Responses at Week 12 | Baseline and Week 12
  Post-stroke fatigue will be assessed using the Fatigue Severity Scale (range: 1-7). Higher scores are indicative of more severe fatigue.
  Health-related quality of life will be assessed using 12-Item Short Form Health Survey (range: 0-100). Higher scores are indicative of better quality of life.
  Exercise enjoyment will be assessed by the Physical Activity Enjoyment Scale and Behavioural Regulation Exercise Questionnaire-3 (range: 0-400). Higher scores indicate a higher exercise enjoyment level.
  Motivation for exercise will be assessed using the Behavioural Regulation Exercise Questionnaire-3 (range: 0-96). Higher scores indicate more motivation to exercise. A semi-structured interview will be additionally conducted at the end of the intervention (week 12) to explore the experiences of HIIT in stroke patients.
  Change=(Week 12 Score - Baseline Score)
Change from Baseline in Psychosocial Responses at Week 24 | Baseline and Week 24
  Post-stroke fatigue will be assessed using the Fatigue Severity Scale (range: 1-7). Higher scores are indicative of more severe fatigue.
  Health-related quality of life will be assessed using 12-Item Short Form Health Survey (range: 0-100). Higher scores are indicative of better quality of life.
  Exercise enjoyment will be assessed by the Physical Activity Enjoyment Scale and Behavioural Regulation Exercise Questionnaire-3 (range: 0-400). Higher scores indicate a higher exercise enjoyment level.
  Motivation for exercise will be assessed using the Behavioural Regulation Exercise Questionnaire-3 (range: 0-96). Higher scores indicate more motivation to exercise. A semi-structured interview will be additionally conducted at the end of the intervention (week 12) to explore the experiences of HIIT in stroke patients.
  Change=(Week 24 Score - Baseline Score)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No